CLINICAL TRIAL: NCT00690885
Title: Evaluation of Natural Human Interferon Alpha Lozenges in the Treatment of Chronic Cough in Patients With Chronic Obstructive Pulmonary Disease (COPD) or Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Interferon-alpha Treatment of Chronic Cough in Chronic Obstructive Pulmonary Disease and Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient patient accrual
Sponsor: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07HUCO01
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Cough
Keywords: chronic cough; COPD; IPF; interferon alpha
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Cough; Chronic Cough | interventions — Interferon-alpha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): lozenges containing 150 IU of natural human interferon-alpha
  Interventions: Drug: interferon-alpha lozenges
- 2 (Placebo Comparator): matching placebo lozenges
  Interventions: Drug: placebo lozenges

INTERVENTIONS:
Drug: interferon-alpha lozenges — 150 IU natural human interferon-alpha lozenges for oral dissolution given 3 times per day for 4 weeks
  Other Names: oral IFN-alpha; oral IFN-alpha lozenges; Veldona lozenges
  Arms: 1
Drug: placebo lozenges — matching placebo lozenges
  Other Names: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether lozenges containing interferon-alpha can reduce the frequency and severity of coughing in patients with chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
Both chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF) frequently lead to a chronic cough that negatively impacts the quality of life (QOL) for patients and those around them. This is a randomized, double-blind, placebo-controlled trial to determine whether interferon-alpha, delivered in low doses via orally dissolving lozenges given 3 times per day for 4 weeks, can reduce the frequency and severity of chronic cough in patients with COPD or IPF. Cough frequency will be assessed via 24-hour digital audio recordings made prior to entry, and at weeks 2 and 4 of treatment. Cough severity will be assessed via a 100-mm visual analog scale questionnaire completed by the subject prior to entry and then weekly during treatment. Subjects will also complete questionnaires regarding cough frequency, duration and intensity, QOL, dyspnea, and antitussive medication usage weekly during treatment. All questionnaires will be repeated weekly during a 4-week post-treatment observation period to assess durability of response.

ELIGIBILITY:
Inclusion Criteria:

For all patients

* history of clinically significant chronic cough for > 3 months
* For COPD patients
* >40 years of age
* 20-pack-year history of smoking
* GOLD classification of Stage 1 or higher
* For IPF patients
* > 50 years of age
* history of unexplained dyspnea on exertion of > 3 months
* exhibits coughing and bilateral, basilar, inspiratory crackles on physical exam
* presents as being in a stable phase of IPF
* lung biopsy or HRCT indicative of IPF

Exclusion Criteria:

* ACE inhibitor use
* GERD
* current cancer or history of lung cancer
* non-ambulatory
* hospitalized in the previous 12 months for heart failure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
frequency/severity of cough | weekly

SECONDARY OUTCOMES:
quality of life | weekly
anti-tussive medication usage | weekly
dyspnea | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz O Lutherer, MD, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Lutherer, LO, et al. Preliminary Results Suggest Prevention of Progression of Idiopathic Pulmonary Fibrosis by Treatment with Low-Dose, Oral Interferon Alpha. Journal of Investigative Medicine 54(1):S278, 2006.
- See also: American Lung Association - COPD fact sheet — http://www.lungusa.org/lung-disease/pulmonary-fibrosis/
- See also: American Lung Association - Interstitial Lung Diseases and Pulmonary Fibrosis — http://www.lungusa.org/lung-disease/copd/